CLINICAL TRIAL: NCT01476059
Title: Prospective, Parallel-group, Randomized Study to Evaluate the Compliance to the Treatment of Children Aged Between 6 and 14 Years Old With Persistent Moderate or Severe Asthma, Receiving the Association Fluticasone 250 mcg/Dose and Salmeterol 50 mcg/Dose Twice a Day. ADERE PROJECT
Brief Title: Pediatric Study to Evaluate Treatment of Persistent Moderate or Severe Asthma With the Association Fluticasone 250 mcg/Dose and Salmeterol 50 mcg/Dose - ADERE PROJECT
Acronym: ADERE (Ped)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113244
Record Dates: First submitted 2010-03-04; First posted 2011-11-22 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: Treatment compliance; Pediatric; Asthma
MeSH Terms: conditions — Asthma; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- telephone follow-up (Other): Asthmatic children being treated, who will be given medical guidance and therapeutic guidance through telephone calls at every fifteen days to the parents or guardians, performed by trained professionals.
  Interventions: Other: Telephone follow-up
- No telephone follow-up (Other): Asthmatic children being treated, who will be given medical guidance without telephone follow-up calls to parents or guardians.
  Interventions: Other: No telephone follow-up

INTERVENTIONS:
Other: Telephone follow-up — Asthmatic children being treated, who will be given medical guidance and therapeutic guidance through telephone calls at every fifteen days to the parents or guardians, performed by trained professionals.
  Arms: telephone follow-up
Other: No telephone follow-up — Asthmatic children being treated, who will be given medical guidance without telephone follow-up calls to parents or guardians.
  Arms: No telephone follow-up

SUMMARY:
Prospective, parallel-group, randomized study to evaluate the compliance to the treatment of children aged between 6 and 14 years old with persistent moderate or severe asthma, receiving the association Fluticasone 250 mcg/dose and Salmeterol 50 mcg/dose twice a day.

ADERE PROJECT (Pediatric)

DETAILED DESCRIPTION:
Objectives

General:

To evaluate the compliance degree to the treatment of asthmatic children, according to the attention received.

Specific:

1. To study asthmatic compliance to the treatment proposed, aiming at an association with other factors, such as: parents' instruction, hospitalizations, personal and family history of atopy, co-morbidities, severity of the disease and use of other drugs.
2. To study asthmatic compliance to the treatment proposed, associating it with the impact in quality of life, though the application of a specific questionnaire.

Outcomes

The main outcome, compliance, is being measured by the number of doses used of the drug salmeterol combined with fluticasone (Seretide Diskus) divided by the number of doses foreseen for the time considered.

The following will be considered as secondary outcomes:

* Disease control, evaluated by information in the questionnaires.
* Regular medical attention sought, evaluated by information in the questionnaires.
* Additional resources in the event of attacks, increase in the weekly number of nocturnal awakening or the number of awakenings per night, increase in the use of rescue drug.
* Improvement in the quality of life.

Casuistic and Method

Study groups

Asthmatic children aged 6 to 14 years old from both sexes, with persistent mild, moderate or sever asthma classified according to the criteria from the III - Brazilian Consensus on Asthma Management.

Group I - Asthmatic children being treated, who will be given medical guidance and therapeutic guidance through telephone calls at every fifteen days to the parents or guardians, performed by trained professionals.

Group II - Asthmatic children being treated, who will be given medical guidance without telephone follow-up calls to parents or guardians.

Study Design

This is a prospective, controlled, randomized, parallel-group study, with the inclusion of 472 children presenting persistent moderate or severe asthma. Our researchers developed the study, and it will be performed only in Brazil, solely by our Clinical Research Center. The drug to be used is in accordance with the main International Consensus on Asthma Treatment and with the III - Brazilian Consensus on Asthma Management, being marketed for some years in Brazil.

During patient recruitment and screening, their parents or guardians will fill out the free informed consent form. At this time, they will also be given the drug (Seretide Diskus® 50/250) with doses enough for a 90-day treatment, twice a day, in addition to instructions on the use of the device to apply the drug and guidance from his/her physician on how to act in the event of an attack.

After study inclusion, the study will receive a number which will randomly include him/her in group 1 or 2 of this study.

Patients included in group 1 will receive two types of telephone calls:

A. Investigation telephone call - TI: that will be made by a trained health professional from the Centro de Pesquisa Clínica e Medicina Avançada, aiming at: presentation, data collection on asthma, including demographics and relevant clinical history (details on asthma, previous exacerbations, drugs used, etc), submission of a standardized checking questionnaire (questionnaire 1 - attachment 1) and quality of life questionnaire (questionnaire 2 - attachment 2). By 90 days, the patient's guardian will receive the last investigation telephone call (TI -2) in order to apply the quality of life questionnaire and standardized evaluation questionnaire (questionnaire 1 - attachment 1)

B. Compliance telephone call - TA: A specifically trained professional will make follow-up telephone calls at every fifteen days, according to a pre-established guide (Attachment 4), requesting the patient to answer the questions pursuant to the follow-up questionnaire (attachment 3) and clarifying probable doubts on the drug application, however, without interfering with the treatment prescribed by the physician.

Patients included in group 2 will receive only the Investigation Telephone call (TI) All telephone contacts will be made for the same person: mother, father or guardian.

By the end of week 12, the persons responsible for the patients will return, by mail, the drug to Centro de Pesquisa Clínica e Medicina Avançada.

ELIGIBILITY:
Inclusion criteria:

* Signature of a informed consent form
* Age between 6 and 14 years old
* Diagnosis of persistent moderate or severe asthma, according to III Brazilian Consensus on Asthma Management.
* Home telephone available

Exclusion criteria:

* Co-morbidities that may interfere with the study evaluation or that require continuous drugs, e.g., cardiopathy, gastro-esophageal reflux or diabetes.
* Continuous systemic corticosteroid use for more than seven days
* The patient has been treated or is being treated with allergen-specific immunetherapy

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 472 (Actual)
Dates: Start 2004-05; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The main outcome, compliance, is being measured by the number of doses used of the drug salmeterol combined with fluticasone (Seretide Diskus) divided by the number of doses foreseen for the time considered. | After 90 days of treatment

SECONDARY OUTCOMES:
Disease control, evaluated by information in the questionnaires. | After 90 days of treatment
Regular medical attention sought, evaluated by information in the questionnaires | After 90 days of treatment
Additional resources in the event of attacks | After 90 days of treatment
Improvement in the quality of life. | After 90 days of treatment
Increase in the weekly number of nocturnal awakening or the number of awakenings per night | After 90 days of treatment
Increase in the use of rescue drug | After 90 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline